CLINICAL TRIAL: NCT05926973
Title: Vector Change Defibrillation in Refractory Shockable Rhythms
Acronym: VOCALIST
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Thames Valley Air Ambulance (Other)
Responsible Party: Principal Investigator, James Raitt, Audit, Improvement and Research Lead, Thames Valley Air Ambulance
Other Study IDs: TVAA02/23
Record Dates: First submitted 2023-05-22; First posted 2023-07-03 (Actual); Last update posted 2023-07-03 (Actual); Status verified 2023-06

CONDITIONS: Cardiac Arrest; Ventricular Fibrillation; Ventricular Tachycardia
Keywords: cardiac arrest; Refractory shockable rhythm; defibrillation
MeSH Terms: conditions — Heart Arrest; Ventricular Fibrillation; Tachycardia, Ventricular

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Before intervention: Standard care as per ALS guidelines prior to October 2021
- After intervention: Enhanced cardiac arrest management as per TVAA guideline from October 2021 onwards
  Interventions: Other: Enhanced cardiac arrest bundle

INTERVENTIONS:
Other: Enhanced cardiac arrest bundle — * Delivering shocks with the LUCAS mechanical CPR device running
  * After 5 shocks have been delivered placing new pads in the Anterior Posterior (AP) position
  * Delivering shocks using the TVAA Tempus Pro defibrillator rather than the Ambulance Service defibrillator.
  Other Names: Vector change defibrillation
  Groups: After intervention

SUMMARY:
Management of cardiac arrest according to published guidelines has remained largely unchanged for a decade. Thames Valley Air Ambulance provide Critical Care Paramedic and Physician teams who respond to cardiac arrests and offer treatments beyond the scope of ambulance service clinicians. Following a review of practice and appraisal of evidence the investigators developed an additional algorithm for cases of adult medical cardiac arrest with refractory shockable rhythms. This adds to but does not replace the Advanced Life Support algorithm and includes:

* Delivering shocks with the LUCAS mechanical CPR device running
* After 5 shocks have been delivered placing new pads in the Anterior Posterior (AP) position
* Delivering shocks using the TVAA Tempus Pro defibrillator rather than the Ambulance Service defibrillator.

This bundle was based on recommendations from ILCOR and the Resus Council (UK) Advanced Life Support manual and was launched in October 2021.

DETAILED DESCRIPTION:
Study hypothesis An enhanced algorithm for refractory shockable rhythms terminates VF/VT and improves outcomes (ROSC at hospital) in out of hospital cardiac arrest.

Study design

PICOST Population - adult patients with medical cardiac arrest in refractory shockable rhythms (defined as continuous VF or VT after 5 shocks).

Intervention - application of the TVAA enhanced cardiac arrest bundle Comparison - 18 month period before the introduction of the bundle (if the COVID period has significantly different response times than the intervention group then the COVID period will be excluded).

Outcome - primary outcome measure is ROSC at hospital (as this represents the success of the pre-hospital phase of resuscitation).

Study design - Retrospective observational study using the TVAA HEMSBASE database Timeframe - 18 months of data since the bundle was introduced.

Exclusions - traumatic cardiac arrests, cardiac arrests where the VF/VT was recurrent (could be terminated but then restarted) rather than refractory (unable to get the patient out of the shockable rhythm). Refractory VF refers to VF that persists despite shock delivery (i.e. shock-resistant VF). This is distinguished from recurrent VF, which is VF that re-appears after it has been terminated (2). In this study refractory would be defined as continuous VF or VT after 5 shocks.

Data set to be collected All data is held within HEMSBASE Age, sex, witnessed arrest, bystander CPR, time from 999 call to TVAA on scene, first rhythm, number of shocks (total in before group; number of shocks pre and post vector change in the after group), outcome (ROSC at any stage; PLE, died on arrival to ED, ROSC in ED).

Statistical analysis Statistical support will be sought from the South Central Research Design Service https://www.rds-sc.nihr.ac.uk Fisher's test or Chi square tests may be appropriate.

Ethical approval The HRA decision tools indicate that the study does not require REC review.

Search strategy Two independent researchers will search HEMSBASE for the intervention period (Oct 21 to April 23) and the control period (19 months prior to Oct 21, excluding the COVID period if response times are significantly different in this period) using the following strategy.

HEMSBASE search

* Cardiac arrests
* Initial rhythm VF or VT
* Manual search looking for refractory shockable rhythms (defined as continuous VF or VT after 5 shocks with no change to ROSC or a non shockable rhythm at any stage).

This search strategy will deliver a list of cases of refractory shockable rhythms that can then be compared between the two reviewers to ensure all cases are included, any cases where there is not agreement will be adjudicated by a third reviewer. The cases will then be analysed for the data set above and entered into an excel spreadsheet.

Data security No patient identifiable data will be exported outside of HEMSBASE.

ELIGIBILITY:
Inclusion Criteria:

* adult patients with medical cardiac arrest
* in refractory shockable rhythms (defined as continuous VF or VT after 5 shocks).

Exclusion Criteria:

* traumatic cardiac arrests
* cardiac arrests where the VF/VT was recurrent (could be terminated but then restarted) rather than refractory (unable to get the patient out of the shockable rhythm). Refractory VF refers to VF that persists despite shock delivery (i.e. shock-resistant VF). This is distinguished from recurrent VF, which is VF that re-appears after it has been terminated (2). In this study refractory would be defined as continuous VF or VT after 5 shocks.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Adult patients with medical cardiac arrest attended by TVAA, in refractory shockable rhythms (defined as continuous VF or VT after 5 shocks).
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2023-05-01 (Actual); Primary Completion 2023-06-30 (Estimated); Study Completion 2023-09 (Estimated)

PRIMARY OUTCOMES:
ROSC at hospital | within 24 hours of arrest
  ROSC at hospital

SECONDARY OUTCOMES:
PLE rate | within 24 hours of arrest
  PLE - death declared at scene

OTHER OUTCOMES:
Total defibrillation shocks | within 24 hours of arrest
  Total defibrillation shocks

CONTACTS AND LOCATIONS:
Locations (1):
- Thames Valley Air Ambulance, Oxford, Oxfordshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No
No individual patient data to be shared